CLINICAL TRIAL: NCT07233382
Title: Assessing the Efficacy of Probiotics in Prevention of NEC in Preterm Babies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hayatabad Medical Complex (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ERB # 2731; Agha Khan (Other Grant/Funding Number: Agha Khan)
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: NEC; NEC - Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Probiotics; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic group - Intervention (Active Comparator): This group will receive intervention
  Interventions: Drug: Probiotic
- Placebo (Placebo Comparator): This group will receive 10% DW
  Interventions: Drug: 10% dextrose

INTERVENTIONS:
Drug: Probiotic — All preterm babies <34 weeks Gestational age admitted within 24 hrs of life will be eligible for the study. Those full filling inclusion criteria and consenting to participate will be recruited. Consent will be obtained by team not caring for the patient. Each recruited patient will be assigned a case ID number. Based on the Randomization babies will be assigned to either the intervention group or control group.
  Study group: Multistrain probiotic containing a mix of Lactobacillus and Bifidobacterium spp.
  * Dose is 1 million international units (0.2ml or 5 drops) OD
  * Started as soon as feed is in initiated
  Other Names: Multistrain Probiotic
  Arms: Probiotic group - Intervention
Drug: 10% dextrose — This will receive 10% DW as placebo
  Other Names: Dextrose water
  Arms: Placebo

SUMMARY:
The goal of the study is to check efficacy of probiotics in preventing necrotizing enterocolitis. The main questions would be if the preterm baby developed NEC or not.

DETAILED DESCRIPTION:
: In the last five years, many systematic reviews have shown the benefit of Probiotics in prevention of NEC and Sepsis in preterm babies but most of these studies have been done in the developed countries. Although the overall benefit has been tilted In favor of use of probiotic however a definitive consensus has not been reached due to inconsistencies in results. Moreover, the impact of multistrain probiotics in our particular population has not been studied, which provides the rationale for our research

ELIGIBILITY:
Inclusion Criteria:

* Male and female preterm infants with a gestational age less than 35 weeks.
* All indoor patients and outdoor patients who present within 24hrs of birth

Exclusion Criteria:

* • Infants with congenital or developmental gastrointestinal disorders for example omphalocele, malrotation, gastroschisis.

  * Infants with severe sepsis or gastrointestinal bleeding on presentation

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 196 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop NEC on probiotic vs placebo | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Romisa Romisa, MBBS, FCPS, Principal Investigator — Hyatabad Medical Complex

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pammi M, Cope J, Tarr PI, Warner BB, Morrow AL, Mai V, Gregory KE, Kroll JS, McMurtry V, Ferris MJ, Engstrand L, Lilja HE, Hollister EB, Versalovic J, Neu J. Intestinal dysbiosis in preterm infants preceding necrotizing enterocolitis: a systematic review and meta-analysis. Microbiome. 2017 Mar 9;5(1):31. doi: 10.1186/s40168-017-0248-8. PMID 28274256